CLINICAL TRIAL: NCT03017183
Title: Detection of Heterogeneity in Central Lung Cancer - Prospective Randomized Controlled Trial to Evaluate the Diagnostic Value of EBUS-TBNA and ctDNA Analysis Compared to Endobronchial Forceps Biopsy
Brief Title: Detection of Heterogeneity in Central Lung Cancer - EBUS-TBNA and ctDNA Analysis vs. Endobronchial Forceps Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wissenschaftliches Institut Bethanien e.V (Other)
Collaborators: AstraZeneca (Industry); Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: WI_EBUS-TBNA_16-226
Record Dates: First submitted 2017-01-05; First posted 2017-01-11 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EBUS-TBNA - Endobrochial Forceps Biopsy (Other): In this arm, EBUS-TBNA will be done first, followed by endobronchial forceps biopsy
  Interventions: Procedure: EBUS-TBNA; Procedure: Endobronchial forceps biopsy
- Forceps - EBUS-TBNA (Other): In this arm, endobronchial forceps biopsy will be done first, followed by EBUS-TBNA
  Interventions: Procedure: EBUS-TBNA; Procedure: Endobronchial forceps biopsy

INTERVENTIONS:
Procedure: EBUS-TBNA — Endobronchial ultrasound guided transbronchial needle aspiration
Procedure: Endobronchial forceps biopsy — Conventional endobronchial forceps biopsy

SUMMARY:
Study participants will be selected from clinical routine patients with endobronchial infiltration of a central lung cancer and indication for bronchoscopic sampling.

Consented patients will undergo bronchoscopy for tumor sampling applying two routine sampling methods during one single procedure (EBUS-TBNA and conventional forceps sampling). The sequence of both sampling methods will be randomized in advance.

The resulting tissue samples will be analyzed by a pathologist using multiplex PCR and FISH. The corresponding analysis results will be compared between sampling methods.

Assignment of a subject to a particular therapeutic strategy is not influenced by this protocol. Medicinal products will be used according to current practice and marketing authorisation.

ELIGIBILITY:
Inclusion criteria:

Subjects eligible for enrolment in the study must meet all of the following criteria:

1. Informed consent: a signed and dated written informed consent prior to study participation.
2. Type of subject: inpatient
3. Age: subjects of more than 18 years and less than 85 years.
4. Central lesion in computed tomography highly suspicious of lung cancer with clinical indication for further diagnostic applying bronchoscopy.
5. Central lesion has to be accessible by the biopsy techniques under investigation

Exclusion criteria:

Subjects meeting any of the following criteria must not be enrolled in the study:

1. Females who are pregnant or lactating , who decide not to undergo a bronchoscopy due to the risk for their child
2. Any contraindication for bronchoscopy and EBUS-TBNA (IBNLT: INR>2, thrombocytopenia <40/nl)
3. Drug/alcohol abuse impairing cognitive knowledge which is needed for a GCP conform informed consent.
4. Inability to read or inability of language: in the opinion of the investigator, any subject who is unable to read and/or would not be able to complete study related materials.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Number of detected mutations | within 7 days after biopsy
  The number of different mutations detected based on each biopsy method as well as ctDNA analysis is determined

CONTACTS AND LOCATIONS:
Overall Officials: Winfried J Randerath, Prof. Dr., Principal Investigator — Wissenschaftliches Institut Bethanien e.V
Locations (1):
- Krankenhaus Bethanien gGmbH, Solingen, North Rhine-Westphalia, Germany